CLINICAL TRIAL: NCT05050357
Title: Effectiveness of Hormonal Intrauterine Device in Treating Pelvic Congestion Syndrome Compared to Oral Progestin
Brief Title: Effectiveness of Hormonal Intrauterine Device in Treating PCS Compared to Oral Progestin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelhamid Mohamed Abdelrahim AboDooh, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIUD vs progestin in PCS
Record Dates: First submitted 2021-07-26; First posted 2021-09-20 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Congestion
Keywords: pelvic congestion syndrome; progestin; Hormonal intrauterine device; Intrauterine system

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hormonal intrauterine device arm (Active Comparator)
  Interventions: Device: Hormonal intrauterine device
- progestin arm (Active Comparator)
  Interventions: Drug: Progestins Norethindrone

INTERVENTIONS:
Device: Hormonal intrauterine device — insertion of hormonal IUD during menstrual period
  Arms: hormonal intrauterine device arm
Drug: Progestins Norethindrone — oral ethisteron twice daily for three months
  Arms: progestin arm

SUMMARY:
The aim of this study is to compare the effectiveness of hormonal intrauterine device (IUD) in treatment of pelvic congestion syndrome in comparison with oral progestins treatment.

DETAILED DESCRIPTION:
Pelvic congestion syndrome (PCS) is a poorly understood association between varicose or dilated pelvic veins and chronic pelvic pain (CPP). It is also called Pelvic venous syndrome, Pelvic venous insufficiency, Pelvic varices and Pelvic vascular dysfunction Chronic pelvic pain is defined as chronic or persistent pain perceived in structures related to the pelvis of either men or women for more than 6 months according to The International Association for the Study of Pain (IASP). In other words, chronic pelvic pain with associated ovarian vein varicosities is termed pelvic congestion syndrome (PCS) and is an important but under-diagnosed condition.

Millions of women worldwide\e may suffer with chronic pelvic pain at some time in their life, and the occurrence may be as high as 39.1%. Chronic pelvic pain may account for 10 to 15% of outpatient gynecologic visits in the United States.The typical age of patients with this condition ranges from 20 to 45 years. It is unclear whether there is any genetic or ethnic predilection.

The etiology of pelvic congestion syndrome is reflux of blood in the ovarian veins due to the absence of functioning valves, resulting in retrograde blood flow and eventual venous dilatation. The cardinal presenting symptom of PCS is pelvic pain, usually described as a dull ache, without evidence of inflammatory disease. Clinical signs may include vulvar varicosities extending onto the medial thigh and long saphenous territory as well as tenderness on deep palpation at the ovarian point; however, such signs are not always present.

For many women with PCS, the road toward a definitive diagnosis has been long and laborious. Certainly the diagnosis of PCS continues to challenge all physicians involved. However, a heightened awareness and clinical suspicion for the specific symptomatology and associated findings may bring about a more rapid progression to the much anticipated treatment. Pelvic ultrasound (US) and/or computed tomography (CT) scan are usually the first imaging modalities in the evaluation of patients with chronic pelvic pain. Both provide excellent resolution of the uterus. Although a CT scan has greater sensitivity for showing varicosities throughout the lower pelvis, Two dimensional ultrasound with Doppler examination provides dynamic information about visualized venous blood flow.

Laparoscopy is often used in patients with chronic pelvic pain in search of a specific diagnosis. This direct visualization is excellent for ruling out other etiologies distinct from PCS such as endometriosis. However, because the examination is done supine and requires insufflation of CO2 gas, there may be compression of varices if present, thereby masking the diagnosis of PCS.Certainly, the diagnostic venogram continues to provide physicians with a reliable minimally invasive gold standard tool in patients with PCS.The diagnostic venogram gives immediate dynamic flow information and measurements of ovarian and pelvic veins with the option of changing patient position.

Many treatment modalities have been proposed. Medical management with hormone analogues and analgesics, surgical ligation of ovarian veins, hysterectomy with or without bilateral salpingo-oophorectomy and transcatheter embolization have been described in the literature as treatment options for patients with PCS today. Medical treatment of PCS includes psychotherapy, progestins, danazol, phlebotonics, gonadotropins receptor agonists (GnRH) with hormone replacement therapy (HRT), dihydroergotamine, and nonsteroidal antiinflammatory drugs (NSAIDS).

To improve clinical efficacy and reduce perioperative and postoperative morbidity, percutaneous pelvic vein embolization therapy has been utilized. Since its introduction in 1993 by Edwards et al, this modality has revolutionized the treatment of PCS. The procedure is usually performed at the time of diagnostic venography using a variety of embolic agents, including sclerosant foam and coils. In several published series in the 1990s, success rates for reduction of chronic pelvic pain ranged from 50 to 80%. With advancements in technique, clinical success is achieved in 70 to 85% of treated patients. It was found taht there was significant improvement in 83% of women in their overall pain perception levels with a mean of 45 months of long-term follow up.

Embolotherapy for PCS is an exciting therapy that has proven to be safer over the past two decades.Chung et al examined the effect of patient stress level on treatment efficacy, directly comparing hysterectomy with oophorectomy versus venous embolization for the treatment of PCS. Analysis of pain scores showed that venous embolization was more effective than hysterectomy, especially for patients who are "typically or moderately highly stressed. It was demonstrated that PCS patients who underwent ovarian and pelvic venous embolization have a more durable result in reduction of their pelvic pain.It was reported that there were no major complications and also did not find any significant changes in the basal follicle-stimulating hormone, luteinizing hormone, or estradiol levels.

Reported complications of embolotherapy are rare (< 4%) and include ovarian vein thrombophlebitis, recurrence of varices, migration of embolic material, and radiation exposure to ovaries. Long-term data shows no demonstrable negative effects on menstrual cycle or fertility from trans-catheter embolotherapy, It has proven to be a safe and effective nonsurgical approach in reducing chronic pelvic pain associated with pelvic venous incompetence.

Regarding this study, investigators hypothesize that levonorgestrel-releasing intrauterine device is better than and more effective than oral progestin in treatment of PCS. Because levonorgestrel-releasing intrauterine device is local treatment and may cause little side effects than the oral treatment. In addition, it has better compliance than oral treatment. Lastly, it contains higher concentration than oral treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical symptoms of pelvic congestion syndrome documented by Trans abdominal and/or transvaginal Doppler ultrasound (dilated ovarian veins with reversed caudal flow, presence of varices , dilated arcuate veins crossing the uterine myometrium, polycystic changes of the ovary and variable duplex waveform during the Valsalva's maneuver).

Exclusion Criteria:

* Endometriosis.
* Uterine fibroids.
* Previous pelvic operations.
* Urological diseases.
* Patient seeking pregnancy
* Pelvic inflammatory diseases
* Congenital uterine malformations

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The effectiveness of hormonal IUD in reducing pain in patient with pelvic congestion syndrome in comparison to oral progestin | two years
  The primary outcome measure is to compare the degree of pain reduction according to pain scale ( where the maximum for the scale will be 10 and means severe pain). The minimum of the score will be one and mean very mild pain to no pain ) in pelvic congestion syndrome cases taking hormonal IUD in comparison to those taking oral progestin.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag, Sohag, Egypt

REFERENCES:
- [Background] Champaneria R, Shah L, Moss J, Gupta JK, Birch J, Middleton LJ, Daniels JP. The relationship between pelvic vein incompetence and chronic pelvic pain in women: systematic reviews of diagnosis and treatment effectiveness. Health Technol Assess. 2016 Jan;20(5):1-108. doi: 10.3310/hta20050. PMID 26789334
- [Background] Chung MH, Huh CY. Comparison of treatments for pelvic congestion syndrome. Tohoku J Exp Med. 2003 Nov;201(3):131-8. doi: 10.1620/tjem.201.131. PMID 14649734
- [Background] Edwards RD, Robertson IR, MacLean AB, Hemingway AP. Case report: pelvic pain syndrome--successful treatment of a case by ovarian vein embolization. Clin Radiol. 1993 Jun;47(6):429-31. doi: 10.1016/s0009-9260(05)81067-0. PMID 8519153
- [Background] Freedman J, Ganeshan A, Crowe PM. Pelvic congestion syndrome: the role of interventional radiology in the treatment of chronic pelvic pain. Postgrad Med J. 2010 Dec;86(1022):704-10. doi: 10.1136/pgmj.2010.099473. PMID 21106807
- [Background] Ganeshan A, Upponi S, Hon LQ, Uthappa MC, Warakaulle DR, Uberoi R. Chronic pelvic pain due to pelvic congestion syndrome: the role of diagnostic and interventional radiology. Cardiovasc Intervent Radiol. 2007 Nov-Dec;30(6):1105-11. doi: 10.1007/s00270-007-9160-0. Epub 2007 Sep 6. PMID 17805925
- [Background] Ignacio EA, Dua R, Sarin S, Harper AS, Yim D, Mathur V, Venbrux AC. Pelvic congestion syndrome: diagnosis and treatment. Semin Intervent Radiol. 2008 Dec;25(4):361-8. doi: 10.1055/s-0028-1102998. PMID 21326577
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Kim HS, Malhotra AD, Rowe PC, Lee JM, Venbrux AC. Embolotherapy for pelvic congestion syndrome: long-term results. J Vasc Interv Radiol. 2006 Feb;17(2 Pt 1):289-97. doi: 10.1097/01.RVI.0000194870.11980.F8. PMID 16517774
- [Background] Maleux G, Stockx L, Wilms G, Marchal G. Ovarian vein embolization for the treatment of pelvic congestion syndrome: long-term technical and clinical results. J Vasc Interv Radiol. 2000 Jul-Aug;11(7):859-64. doi: 10.1016/s1051-0443(07)61801-6. PMID 10928522
- [Background] Park SJ, Lim JW, Ko YT, Lee DH, Yoon Y, Oh JH, Lee HK, Huh CY. Diagnosis of pelvic congestion syndrome using transabdominal and transvaginal sonography. AJR Am J Roentgenol. 2004 Mar;182(3):683-8. doi: 10.2214/ajr.182.3.1820683. PMID 14975970
- [Background] Robinson JC. Chronic pelvic pain. Curr Opin Obstet Gynecol. 1993 Dec;5(6):740-3. PMID 8286684
- [Background] Soysal ME, Soysal S, Vicdan K, Ozer S. A randomized controlled trial of goserelin and medroxyprogesterone acetate in the treatment of pelvic congestion. Hum Reprod. 2001 May;16(5):931-9. doi: 10.1093/humrep/16.5.931. PMID 11331640
- [Background] Venbrux AC, Chang AH, Kim HS, Montague BJ, Hebert JB, Arepally A, Rowe PC, Barron DF, Lambert D, Robinson JC. Pelvic congestion syndrome (pelvic venous incompetence): impact of ovarian and internal iliac vein embolotherapy on menstrual cycle and chronic pelvic pain. J Vasc Interv Radiol. 2002 Feb;13(2 Pt 1):171-8. doi: 10.1016/s1051-0443(07)61935-6. PMID 11830623
- [Background] Venbrux AC, Lambert DL. Embolization of the ovarian veins as a treatment for patients with chronic pelvic pain caused by pelvic venous incompetence (pelvic congestion syndrome). Curr Opin Obstet Gynecol. 1999 Aug;11(4):395-9. doi: 10.1097/00001703-199908000-00006. PMID 10498026